CLINICAL TRIAL: NCT00863655
Title: A Randomized Double-Blind, Placebo-Controlled Study of Everolimus in Combination With Exemestane in the Treatment of Postmenopausal Women With Estrogen Receptor Positive Locally Advanced or Metastatic Breast Cancer Who Are Refractory to Letrozole or Anastrozole
Brief Title: Everolimus in Combination With Exemestane in the Treatment of Postmenopausal Women With Estrogen Receptor Positive Locally Advanced or Metastatic Breast Cancer Who Are Refractory to Letrozole or Anastrozole
Acronym: BOLERO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001Y2301; 2008-008698-69 (EudraCT Number)
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Estrogen Receptor positive; ER+; exemestane; mTOR; everolimus; refractory; NSAI
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus + Exemestane (Experimental): Everolimus 10 mg daily in combination with exemestane 25 mg daily
  Interventions: Drug: Everolimus; Drug: Exemestane
- Placebo + Exemestane (Active Comparator): Placebo of everolimus in combination with exemestane 25 mg daily
  Interventions: Drug: Exemestane; Drug: Everolimus Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus was formulated as tablets of 5-mg strength and was packaged into blister packs . Everolimus (two 5 mg tablets daily) were administered in a blinded manner on their respective treatment arms by continuous oral daily dosing.
  Other Names: RAD001
  Arms: Everolimus + Exemestane
Drug: Exemestane — Exemestane 25 mg orally daily.
Drug: Everolimus Placebo — Placebo was formulated to be indistinguishable from the everolimus tablets. Matching placebo (two tablets daily) were administered in a blinded manner on their respective treatment arms by continuous oral daily dosing.
  Arms: Placebo + Exemestane

SUMMARY:
There are no treatments specifically approved after recurrence or progression on a non steroidal aromatase inhibitors (NSAI). In light of the need for new treatment options for postmenopausal women after failure of prior NSAI therapy, the purpose of this Phase III study is to compare efficacy and safety of a treatment with exemestane + everolimus to exemestane + placebo in postmenopausal women with estrogen receptor positive locally advanced or metastatic breast cancer refractory to NSAI.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Histological or cytological confirmation of estrogen-receptor positive (ER+) breast cancer
* Postmenopausal women.
* Disease refractory to non steroidal aromatase inhibitors (NSAI),
* Radiological or clinical evidence of recurrence or progression on or after the last systemic therapy prior to randomization.
* Patients must have at least one lesion that can be accurately measured or bone lesions in the absence of measurable disease as defined above.

Exclusion Criteria:

* HER2-overexpressing patients
* Patients with only non-measurable lesions other than bone metastasis (e.g. pleural effusion, ascites etc.).
* Patients who received more than one chemotherapy line for Advanced Breast Cancer.
* Previous treatment with exemestane or mTOR inhibitors.
* Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin).
* Radiotherapy within four weeks prior to randomization
* Currently receiving hormone replacement therapy,

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2014-12-04 (Actual); Study Completion 2014-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (187):
- United States (63):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Highlands Oncology Group DeptofHighlandsOncologyGrp(2), Fayetteville, Arkansas
  - Kaiser Permanente Medical Group Kaiser Permanente-Moanalua M.C, Anaheim, California
  - Comprehensive Blood and Cancer Center Dept. of CBCC (3), Bakersfield, California
  - Cancer Care Associates Dept.ofCancerCareAssoc. (2), Fresno, California
  - Grass Valley Hematology Oncology Medical Group Dept. of Grass Valley Hem/Onc, Grass Valley, California
  - Scripps Clinic SC, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC/Kenneth Norris Comprehensive Cancer Center Regulatory Contact 3, Los Angeles, California
  - Sharp Memorial Hospital SharpClinicalOncologyResearch, San Diego, California
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - Premiere Oncology/Pinnacle Oncology Hematology Dept.ofPremiereOncologyAZ, Santa Monica, California
  - St Joseph Heritage Healthcare Dept. of RRMG (4), Santa Rosa, California
  - Comprehensive Cancer Center - Boca Raton Deerfield Beach, Boca Raton, Florida
  - Florida Cancer Research Institute, Davie, Florida
  - Florida Cancer Specialists DeptofFloridaCancerSpecialists, Fort Myers, Florida
  - Memorial Hospital Memorial Cancer Institute, Hollywood, Florida
  - MD Anderson Cancer Center - Orlando Dept.ofMDACC-Orlando(2), Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Florida Medical Clinic PA Dept.ofFloridaMedicalClinic, Zephyrhills, Florida
  - Georgia Cancer Specialists. Drug Ship, Decatur, Georgia
  - Rush University Medical Center Study Coordinator, Chicago, Illinois
  - Oncology Specialists, SC Dept.of Oncology Specialists, Park Ridge, Illinois
  - Hematology Oncology of Indiana, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Cancer Center of Kansas Dept.ofCancerCtr.ofKansas, Wichita, Kansas
  - University of Louisville / James Graham Brown Cancer Center SC, Louisville, Kentucky
  - Hematology Oncology Clinic Hematology Oncology Clinic (2), Baton Rouge, Louisiana
  - Crescent City Research Consortium, LLC Dept of Hem&Onc Specialist - 2, Metairie, Louisiana
  - Anne Arundel Health System Research Institute Wayson Pavilion, Annapolis, Maryland
  - Mercy Medical Center Medical Oncology & Hematology, Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square Hospital, Baltimore, Maryland
  - Maryland Hematology/Oncology Associates, P.A., Baltimore, Maryland
  - Frederick Memorial Hospital Dept. of FMH-IRB, Frederick, Maryland
  - Holy Cross Hospital Holy Cross, Silver Spring, Maryland
  - Lahey Clinic Dept of Lahey Clinic (2), Burlington, Massachusetts
  - Fairview Southdale Medical Oncology Clinic, Edina, Minnesota
  - St. Louis Cancer & Breast Institute Dept.ofSt.LouisCancer&Breast, St Louis, Missouri
  - Southeast Nebraska Oncology Cancer Center, Lincoln, Nebraska
  - Regional Cancer Care Associates Dept. of the CCHD, Cherry Hill, New Jersey
  - Trinitas Comprehensive Cancer Center Dept. of Trinitas, Elizabeth, New Jersey
  - University of New Mexico Cancer Research Center Dept of UNM Cancer & Research, Albuquerque, New Mexico
  - Clinical Research Alliance Dept.ofArenaOncologyAssoc(2), Lake Success, New York
  - ProHealth Care, Lake Success, New York
  - Beth Israel Medical Center Dept.ofBeth Israel Med. Ctr(2), New York, New York
  - Weill Cornell Medical College Weill Cornell Med. Ctr., New York, New York
  - Hematology Oncology Association of Rockland, Nyack, New York
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Cancer Centers of Southwest Oklahoma Cancer Research Dept.of Southwest Oklahoma, Lawton, Oklahoma
  - Cancer Care Associates SC, Tulsa, Oklahoma
  - Penn State University / Milton S. Hershey Medical Center Division of Oncology (2), Hershey, Pennsylvania
  - Medical University of South Carolina -Hollings Cancer Center Dept. MUSC/HollingsCancerCtr, Charleston, South Carolina
  - Sarah Cannon Research Institute Dept.ofSarahCannonCancerCtr(5), Nashville, Tennessee
  - University of Texas Southwestern Medical Center SimmonsComprehensiveCancerCtr., Dallas, Texas
  - The Center for Cancer and Blood Disorders Dept. of The Ctr for C & BD(2), Fort Worth, Texas
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(2), Houston, Texas
  - Hope Oncology HOPE Richardson, Richardson, Texas
  - Northern Utah Cancer Associates SC, Ogden, Utah
  - Central Utah Clinic CRAD001Y2301, Provo, Utah
  - Utah Cancer Specialists Dept.of Utah Cancer Spec. (2), Salt Lake City, Utah
  - University of Utah / Huntsman Cancer Institute Dept.ofHuntsmanCancerInst.(2), Salt Lake City, Utah
  - Medical Oncology & Hematology Associates of Northern VA Med. Onc&Hem Assoc. of No.VA, Reston, Virginia
  - University of Wisconsin Hospital & Clinics UW ComprehensiveCancerCtr(2), Madison, Wisconsin
- Australia (5):
  - Novartis Investigative Site, Nambour, Queensland
  - Novartis Investigative Site, Redcliffe, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Subiaco, Western Australia
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Austria
  - Novartis Investigative Site, Wels, Austria
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Sint-Niklaas
  - Novartis Investigative Site, Wilrijk
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (13):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, St. Catharines, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Czechia (3):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
- Egypt (3):
  - Novartis Investigative Site, Menoufiya, Egypt
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- France (8):
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Saint-Nazaire
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Trier
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szolnok
- Italy (10):
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Antella - Bagno A Ripoli, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Saronno, Va
  - Novartis Investigative Site, Varese, VA
- Japan (18):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
- Netherlands (6):
  - Novartis Investigative Site, Eindhoven, Netherlands
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, The Hague
- Novartis Investigative Site, Christchurch, Christchurch, New Zealand
- Novartis Investigative Site, Lørenskog, Norway
- Poland (3):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- South Korea (3):
  - Novartis Investigative Site, Hwasun-gun, Jeollanam-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (10):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
- Sweden (2):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Ankara
- United Kingdom (6):
  - Novartis Investigative Site, Broomfield, Chelmsford
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- [Derived] Chandarlapaty S, Chen D, He W, Sung P, Samoila A, You D, Bhatt T, Patel P, Voi M, Gnant M, Hortobagyi G, Baselga J, Moynahan ME. Prevalence of ESR1 Mutations in Cell-Free DNA and Outcomes in Metastatic Breast Cancer: A Secondary Analysis of the BOLERO-2 Clinical Trial. JAMA Oncol. 2016 Oct 1;2(10):1310-1315. doi: 10.1001/jamaoncol.2016.1279. PMID 27532364
- [Derived] Hortobagyi GN, Chen D, Piccart M, Rugo HS, Burris HA 3rd, Pritchard KI, Campone M, Noguchi S, Perez AT, Deleu I, Shtivelband M, Masuda N, Dakhil S, Anderson I, Robinson DM, He W, Garg A, McDonald ER 3rd, Bitter H, Huang A, Taran T, Bachelot T, Lebrun F, Lebwohl D, Baselga J. Correlative Analysis of Genetic Alterations and Everolimus Benefit in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Results From BOLERO-2. J Clin Oncol. 2016 Feb 10;34(5):419-26. doi: 10.1200/JCO.2014.60.1971. Epub 2015 Oct 26. PMID 26503204
- [Derived] Piccart M, Hortobagyi GN, Campone M, Pritchard KI, Lebrun F, Ito Y, Noguchi S, Perez A, Rugo HS, Deleu I, Burris HA 3rd, Provencher L, Neven P, Gnant M, Shtivelband M, Wu C, Fan J, Feng W, Taran T, Baselga J. Everolimus plus exemestane for hormone-receptor-positive, human epidermal growth factor receptor-2-negative advanced breast cancer: overall survival results from BOLERO-2dagger. Ann Oncol. 2014 Dec;25(12):2357-2362. doi: 10.1093/annonc/mdu456. Epub 2014 Sep 17. PMID 25231953
- [Derived] Rugo HS, Pritchard KI, Gnant M, Noguchi S, Piccart M, Hortobagyi G, Baselga J, Perez A, Geberth M, Csoszi T, Chouinard E, Srimuninnimit V, Puttawibul P, Eakle J, Feng W, Bauly H, El-Hashimy M, Taran T, Burris HA 3rd. Incidence and time course of everolimus-related adverse events in postmenopausal women with hormone receptor-positive advanced breast cancer: insights from BOLERO-2. Ann Oncol. 2014 Apr;25(4):808-815. doi: 10.1093/annonc/mdu009. Epub 2014 Mar 10. PMID 24615500
- [Derived] Yardley DA, Noguchi S, Pritchard KI, Burris HA 3rd, Baselga J, Gnant M, Hortobagyi GN, Campone M, Pistilli B, Piccart M, Melichar B, Petrakova K, Arena FP, Erdkamp F, Harb WA, Feng W, Cahana A, Taran T, Lebwohl D, Rugo HS. Everolimus plus exemestane in postmenopausal patients with HR(+) breast cancer: BOLERO-2 final progression-free survival analysis. Adv Ther. 2013 Oct;30(10):870-84. doi: 10.1007/s12325-013-0060-1. Epub 2013 Oct 25. PMID 24158787
- [Derived] Campone M, Beck JT, Gnant M, Neven P, Pritchard KI, Bachelot T, Provencher L, Rugo HS, Piccart M, Hortobagyi GN, Nunzi M, Heng DY, Baselga J, Komorowski A, Noguchi S, Horiguchi J, Bennett L, Ziemiecki R, Zhang J, Cahana A, Taran T, Sahmoud T, Burris HA 3rd. Health-related quality of life and disease symptoms in postmenopausal women with HR(+), HER2(-) advanced breast cancer treated with everolimus plus exemestane versus exemestane monotherapy. Curr Med Res Opin. 2013 Nov;29(11):1463-73. doi: 10.1185/03007995.2013.836078. Epub 2013 Sep 4. PMID 23962028
- [Derived] Noguchi S, Masuda N, Iwata H, Mukai H, Horiguchi J, Puttawibul P, Srimuninnimit V, Tokuda Y, Kuroi K, Iwase H, Inaji H, Ohsumi S, Noh WC, Nakayama T, Ohno S, Rai Y, Park BW, Panneerselvam A, El-Hashimy M, Taran T, Sahmoud T, Ito Y. Efficacy of everolimus with exemestane versus exemestane alone in Asian patients with HER2-negative, hormone-receptor-positive breast cancer in BOLERO-2. Breast Cancer. 2014 Nov;21(6):703-14. doi: 10.1007/s12282-013-0444-8. Epub 2013 Feb 13. PMID 23404211
- [Derived] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 724 patients were randomized, 4 never received any study treatment and thus were excluded form the safety set.
Period: Overall Study
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Started | 485 | 239
Completed | 0 (Completed means discontinued the treatment period.) | 0 (Completed means discontinued the treatment period.)
Not Completed | 485 | 239
Not completed — Protocol Violation | 4 | 0
Not completed — Adverse Event | 52 | 8
Not completed — Withdrawal by Subject | 47 | 7
Not completed — Administrative problems | 1 | 0
Not completed — Death | 7 | 1
Not completed — New cancer therapy | 5 | 1
Not completed — Disease progression | 364 | 221
Not completed — Treatment completed as per protocol | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane | Total
Number analyzed (Participants) | 485 | 239 | 724
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.31) | 61.2 (9.75) | 62.1 (10.14)
Age, Customized [Number; unit: Participants]
  < 65 years | 290 | 159 | 449
  >= 65 years | 195 | 80 | 275
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 485 | 239 | 724
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Local Radiology Review of Tumor Assessments.
Description: Progression-free survival, the primary endpoint in this study, is defined as the time from the date of randomization to the date of first documented radiological progression or death due to any cause. Disease progression was based on the tumor assessment by the local radiologist or investigator using RECIST 1.0 criteria. If a patient did not progress or known to have died at the date of the analysis cut-off or start of another antineoplastic therapy, the PFS date was censored to the date of last adequate tumor assessment prior to cut-off date or start of antineoplastic therapy. For patients with lytic or mixed (lytic+sclerotic) bone lesions, the following is considered progression: appearance of ≥1 new lytic lesions in bone; the appearance of ≥ new lesions outside of bone and unequivocal progression of existing bone lesions.
Time Frame: date of randomization to the date of first documented tumor progression or death from any cause, whichever occurs first, reported between day of first patient randomized up to about 19 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
months | 6.93 [6.44 to 8.05] | 2.83 [2.76 to 4.14]
Statistical Analysis 1: Comparison: Everolimus + Exemestane vs Placebo + Exemestane; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.35 to 0.54]

2. Secondary Outcome: Overall Survival (OS) by Number of Deaths
Description: Overall survival, the key secondary endpoint in this study, is defined as the time from date of randomization to the date of death due to any cause. If a patient is not known to have died, survival was censored at the date of last contact.
Time Frame: up to 53 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Participants | 267 | 143

3. Secondary Outcome: Overall Survival (OS) by Median
Description: Overall survival, the key secondary endpoint in this study, is defined as the time from date of randomization to the date of death due to any cause.
Time Frame: up to 53 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Months | 30.98 [27.96 to 34.56] | 26.55 [22.57 to 33.08]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) is the percentage of patients with a best overall response of complete response (CR) or partial response (PR) according to RECIST 1.0. Per RECIST criteria 1.0, CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: up to 21 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Percentage of participants | 9.5 | 0.4

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of patients with best overall response of either complete response (CR), a partial response (PR) or stable disease (SD) >= 24 weeks, according to RECIST 1.0. Per RECIST criteria 1.0, CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD; PD = At least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline.
Time Frame: up to 21 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Percentage of participants | 33.4 | 18.0

6. Secondary Outcome: Proportion of Patients With no Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) Using Kaplan-Meier
Description: The ECOG PS (Eastern Cooperative Oncology Group Performance Scale) is a standard criteria for measuring how treatment of cancer impacts level of functioning in terms of the ability to care for oneself, daily activity, & physical ability (walking, working, etc.). Scale score ranges:0 to 5, 5 being the worst. Scale index: 0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature. 2: Ambulatory & capable of all self-care but unable to carry out any work activities. Up & about more than 50% of waking hours. 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. 5 - Dead. A deterioration of ECOG is an increase of 1 of the ECOG PS without improvement back to initial level at a subsequent time of measurement.
Time Frame: 2, 4, 6, 9 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Proportion of patients
  2 Months | 0.84 [0.80 to 0.87] | 0.87 [0.82 to 0.91]
  4 Months | 0.74 [0.70 to 0.78] | 0.80 [0.73 to 0.85]
  6 Months | 0.64 [0.58 to 0.69] | 0.67 [0.57 to 0.75]
  9 Months | 0.57 [0.50 to 0.63] | 0.47 [0.32 to 0.61]

7. Secondary Outcome: Patient-reported Outcomes (PROs): Time to Deterioration of PRO Scores Using Kaplan Meier - EORTC QLQ-C30
Description: The QLQ-C30 is composed of both multi-item scales and single-item measures. These include 5 functional scales, 3 symptom scales, a global health status - QoL scale, and 6 single items. Each of the multi-item scales includes a different set of items - no item occurs in more than 1 scale. All of the scales measures range in score from 0 to 100. A high scale score = higher response level. Thus a high score for a functional scale represents a healthy level of function, a high score for the global health status / QoL represents a high quality of life but a high score for a symptom scale / item represents a high level of symptomatology / problems. The principle for scoring these scales: 1.) Estimate the average of the items that contribute to the scale = raw score. 2.) Linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Time Frame: Up to 21 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Months
  Deterioration global health status score ≥ 5% | 4.53 [4.17 to 5.68] | 4.40 [3.58 to 5.85]
  Deterioration in PF domain score of ≥ 5% | 4.83 [4.17 to 6.97] | 4.37 [2.83 to 7.00]
  Deterioration in EF domain score of ≥ 5% | 6.93 [5.55 to 8.41] | 6.93 [4.17 to 7.36]
  Deterioration in SF domain score of ≥ 5% | 8.34 [6.93 to 10.87] | 7.03 [5.62 to NA] — NA: Median time to definitive deterioration computed using Kaplan-Meier method.95% CIs calculated using Brookmeyer & Crowley (1982) method. Therefore, upper boundary of 95% CI may not be estimable when median is close to the longest patient follow-up

8. Secondary Outcome: Proportion of Patients With Having no Overall Response Based on Investigator Assessment
Description: overall response = complete response (CR) + partial response (PR) per RECIST 1.0 Time to overall response (CR or PR) based on investigator is the time between date of randomization/start of treatment until first documented response (CR or PR). This analysis included all patients/responders. Patients who did not achieve a confirmed PR or CR were censored at last adequate tumor assessment date when they did not progress. Per RECIST criteria 1.0, CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: 2, 4, 6, 9 months
Population: All randomized patients were included in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 485 | 239
Proportion of patients
  2 months | 0.96 [0.94 to 0.98] | 1.00 [0.97 to 1.00]
  4 months | 0.93 [0.91 to 0.95] | 1.00 [0.97 to 1.00]
  6 months | 0.92 [0.89 to 0.94] | 1.00 [0.97 to 1.00]
  9 months | 0.90 [0.88 to 0.93] | 1.00 [0.97 to 1.00]

9. Secondary Outcome: Duration of Response (Among Participants With Best Overall Response of CR or PR) Estimated Per Kaplan-Meier
Description: Duration of response of CR or PR based on investigator applies only to patients whose best overall response was CR or PR (RECIST 1.0). The start date was the date of first documented response (CR or PR) and the end date and censoring is defined the same as that for time to progression. Per RECIST criteria 1.0, CR: Disappearance of all target lesions; PR: At least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: 21 months
Population: Randomized patients with best overall response of CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 46 | 1
Months | 8.21 [5.55 to NA] — NA - upper limit was not estimable | NA [NA to NA] — NA - median, lower and upper limit of the 95 % CI were not estimable

10. Secondary Outcome: Everolimus Concentrations at Week 4
Description: Characterize the pharmacokinetics (PK) of everolimus in combination with exemestane using Cmin (pre-dose) and C2h (post-dose) at week 4 in a small group of patients.
Time Frame: pre-dose, 2 hours post-dose
Population: Safety Set population consisted of all patients who received at least one dose of study treatment and who had at least one valid post-baseline safety assessment. Although the safety set was considered for the analysis (N), only participants (n) who had pre-dose & 2 hours post-dose values for the given time points were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus + Exemestane
Number analyzed (Participants) | 24
ng/mL
  Pre-dose (Cmin) (n:22) | 16.04 (9.356)
  2 hours post-dose (C2h) (n:24) | 46.50 (17.954)

11. Secondary Outcome: Exemestane Concentrations at Week 4
Description: Characterize the PK of exemestane in combination with or without everolimus using Cmin and C2h at week 4 in a small group of patients.
Time Frame: predose, 2 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 39 | 22
ng/mL
  Pre-dose (Cmin) (n: 34, n: 22) | 0.63 (0.474) [1.00 to 1.00] | 0.43 (0.376) [NA to NA]
  2 hours post-dose (C2h) (n: 39, n: 22) | 23.16 (19.805) [0.68 to 0.94] | 13.30 (11.889) [NA to NA]

12. Secondary Outcome: Estradiol Plasma Concentrations
Description: Compare estradiol concentrations from baseline to week 4 in both treatment arms.
Time Frame: Baseline, Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 41 | 15
pg/mL
  Baseline (n: = 41, 14) | 5.62 (3.342) [1.00 to 1.00] | 4.09 (1.792) [NA to NA]
  Week 4 (n: 38, 15) | 3.50 (2.551) [0.68 to 0.94] | 5.17 (6.919) [NA to NA]

ADVERSE EVENTS:
Description: 4 patients were excluded from the Safety Set; all 4 of these patients (3 in the everolimus plus exemestane arm and 1 in the placebo plus exemestane group) were randomized but subsequently didn't receive study treatment and didn't have an AE reported.
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Serious Adverse Events (participants affected / at risk) | 158/482 | 37/238
Other Adverse Events (participants affected / at risk) | 479/482 | 209/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane (N=482) | Placebo + Exemestane (N=238)
Anaemia (Blood and lymphatic system disorders) | 7 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Periodontitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 5 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 4 | 0
Hyperpyrexia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 6 | 4
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 2
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 1 | 0
Computerised tomogram abnormal (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 5 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 3 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Preventive surgery (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 3 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3
Asthenia (General disorders) | 6 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 6 | 0
Hyperpyrexia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 7 | 4
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 3 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0
Groin abscess (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Histoplasmosis (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 3 | 0
Pyometra (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 5 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 0
Renal impairment (Renal and urinary disorders) | 3 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Preventive surgery (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Intra-abdominal haematoma (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 4 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane (N=482) | Placebo + Exemestane (N=238)
Anaemia (Blood and lymphatic system disorders) | 93 | 9
Leukopenia (Blood and lymphatic system disorders) | 27 | 3
Neutropenia (Blood and lymphatic system disorders) | 39 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 61 | 1
Abdominal pain upper (Gastrointestinal disorders) | 34 | 7
Constipation (Gastrointestinal disorders) | 67 | 31
Diarrhoea (Gastrointestinal disorders) | 157 | 44
Dry mouth (Gastrointestinal disorders) | 51 | 16
Nausea (Gastrointestinal disorders) | 138 | 65
Stomatitis (Gastrointestinal disorders) | 281 | 26
Vomiting (Gastrointestinal disorders) | 75 | 27
Asthenia (General disorders) | 63 | 9
Fatigue (General disorders) | 170 | 65
Oedema peripheral (General disorders) | 92 | 15
Pyrexia (General disorders) | 70 | 12
Nasopharyngitis (Infections and infestations) | 46 | 21
Urinary tract infection (Infections and infestations) | 45 | 5
Alanine aminotransferase increased (Investigations) | 57 | 10
Aspartate aminotransferase increased (Investigations) | 64 | 13
Blood alkaline phosphatase increased (Investigations) | 12 | 12
Blood creatinine increased (Investigations) | 36 | 2
Blood lactate dehydrogenase increased (Investigations) | 27 | 4
Gamma-glutamyltransferase increased (Investigations) | 43 | 20
Weight decreased (Investigations) | 119 | 15
Decreased appetite (Metabolism and nutrition disorders) | 142 | 28
Hypercholesterolaemia (Metabolism and nutrition disorders) | 44 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 63 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 26 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 93 | 40
Back pain (Musculoskeletal and connective tissue disorders) | 64 | 23
Bone pain (Musculoskeletal and connective tissue disorders) | 31 | 20
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 29 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 | 25
Dizziness (Nervous system disorders) | 32 | 15
Dysgeusia (Nervous system disorders) | 104 | 14
Headache (Nervous system disorders) | 103 | 34
Insomnia (Psychiatric disorders) | 65 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 116 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 93 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 83 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 26 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 66 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 49 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 35 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 38 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 63 | 11
Rash (Skin and subcutaneous tissue disorders) | 186 | 15
Hot flush (Vascular disorders) | 27 | 34
Hypertension (Vascular disorders) | 39 | 8
Lymphoedema (Vascular disorders) | 25 | 4
Anaemia (Blood and lymphatic system disorders) | 101 | 11
Leukopenia (Blood and lymphatic system disorders) | 29 | 4
Neutropenia (Blood and lymphatic system disorders) | 40 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 63 | 1
Abdominal pain (Gastrointestinal disorders) | 25 | 11
Abdominal pain upper (Gastrointestinal disorders) | 39 | 7
Constipation (Gastrointestinal disorders) | 74 | 31
Diarrhoea (Gastrointestinal disorders) | 172 | 44
Dry mouth (Gastrointestinal disorders) | 55 | 17
Dyspepsia (Gastrointestinal disorders) | 29 | 12
Nausea (Gastrointestinal disorders) | 157 | 69
Stomatitis (Gastrointestinal disorders) | 286 | 28
Vomiting (Gastrointestinal disorders) | 88 | 30
Asthenia (General disorders) | 70 | 11
Fatigue (General disorders) | 180 | 65
Oedema peripheral (General disorders) | 103 | 15
Pyrexia (General disorders) | 82 | 13
Nasopharyngitis (Infections and infestations) | 53 | 21
Upper respiratory tract infection (Infections and infestations) | 32 | 6
Urinary tract infection (Infections and infestations) | 49 | 5
Alanine aminotransferase increased (Investigations) | 66 | 11
Aspartate aminotransferase increased (Investigations) | 75 | 13
Blood alkaline phosphatase increased (Investigations) | 18 | 12
Blood creatinine increased (Investigations) | 41 | 3
Blood lactate dehydrogenase increased (Investigations) | 30 | 4
Gamma-glutamyltransferase increased (Investigations) | 53 | 20
Weight decreased (Investigations) | 136 | 17
Decreased appetite (Metabolism and nutrition disorders) | 148 | 31
Hypercholesterolaemia (Metabolism and nutrition disorders) | 50 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 69 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 29 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 39 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 107 | 41
Back pain (Musculoskeletal and connective tissue disorders) | 81 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 31 | 15
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 38 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 30 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 35 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 | 26
Dizziness (Nervous system disorders) | 38 | 16
Dysgeusia (Nervous system disorders) | 106 | 14
Headache (Nervous system disorders) | 112 | 35
Anxiety (Psychiatric disorders) | 25 | 6
Depression (Psychiatric disorders) | 28 | 11
Insomnia (Psychiatric disorders) | 68 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 129 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 105 | 25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 86 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 73 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 51 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 39 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 40 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 64 | 11
Rash (Skin and subcutaneous tissue disorders) | 190 | 16
Hot flush (Vascular disorders) | 31 | 34
Hypertension (Vascular disorders) | 49 | 9
Lymphoedema (Vascular disorders) | 30 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data in the clinical trial.